CLINICAL TRIAL: NCT00812305
Title: A Randomized, Double-Blind, Phase 1 Study to Assess the Pharmacokinetics and Safety of SKY0402 in Subjects With Impaired Hepatic Function
Brief Title: Hepatic Impairment Study: Pharmacokinetics in Healthy and Hepatically Impaired Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Ronald M. Burch, MD, PhD, CMO, Pacira Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKY0402C110
Record Dates: First submitted 2008-12-09; First posted 2008-12-22 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Pain; Hepatic Impairment
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose in healthy patients (Experimental)
  Interventions: Drug: SKY0402 300mg in healthy patients
- Low dose in hepatically impaired patients (Experimental)
  Interventions: Drug: SKY0402 300mg in hepatically impaired patients

INTERVENTIONS:
Drug: SKY0402 300mg in healthy patients — SKY0402, single administration of 300 mg via local infiltrations (subcutaneous) in healthy patients
  Other Names: Healthy and Hepatic Impaired subjects will receive SKY0402.
  Arms: Low dose in healthy patients
Drug: SKY0402 300mg in hepatically impaired patients — SKY0402, single administration of 300 mg via local infiltrations (subcutaneous) in hepatically impaired patients
  Other Names: Healthy and Hepatic Impaired subjects will receive SKY0402.
  Arms: Low dose in hepatically impaired patients

SUMMARY:
Review differences between how a healthy person and how a person with liver problems handles the study drug.

DETAILED DESCRIPTION:
Evaluate the pharmacokinetic (PK) profile of SKY0402 in subjects with moderate hepatic impairment compared with age-, gender-, and weight-matched control subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

All Subjects:

* Male or female, ages 18-65 years, inclusive, at Screening. Eligible female subjects of childbearing potential with a nonsterilized male sexual partner must agree to use a hormonal contraceptive, barrier contraceptive with additional spermicide, or an intrauterine device beginning >30 days prior to study drug administration and continuing until >7 days after the end of the study. Female subjects who are postmenopausal must have been postmenopausal for >1 year if they wish not to use contraceptives. If postmenopausal status is questionable, the subject's follicle stimulating hormone (FSH) level must be checked and must be elevated and consistent with postmenopausal levels (i.e., >40 IU/L); otherwise these subjects must agree to use contraceptives listed above.
* Able and willing to comply with all study visits and procedures, including returning as scheduled for post-treatment visits.
* Able to speak, read, and understand the language of the informed consent, and any other instruments used for collecting subject-reported outcomes, in order to enable accurate and appropriate responses to study assessments.
* Willing and capable of providing written informed consent.

Subjects with Hepatic Impairment:

* Subjects must have a positive diagnosis of liver cirrhosis (hepatic fibrosis with evidence of either micro- or macro-nodular regeneration) that has been stable for two months and is confirmed by imaging techniques, biopsy, or physical signs consistent with a clinical diagnosis of liver cirrhosis (e.g., liver firmness to palpation, splenic enlargement, spider angiomata, palmar erythema, parotid hypertrophy, testicular atrophy, gynecomastia).
* Subjects must have an impaired but stable hepatic function evidenced by Child-Pugh Clinical Assessment Score between 7 and 9 at both screening and baseline.

Control Subjects with Normal Hepatic Function:

* Subjects must be in general good health as determined by past medical history, physical examination, vital signs, electrocardiogram, Chest X-Ray (CXR), and laboratory tests at screening.
* Subjects should be matched to a hepatically impaired subject in gender, age (±15%) and weight (±20%).

Exclusion Criteria:

All Subjects

* A history of hypersensitivity to amide type local anesthetics.
* Pregnancy, nursing, or planning to become pregnant during the course of the study.
* Body weight less than 60 kg (~132 lbs) or more than 120 kg (~264 lbs).
* BMI of less than 18 or more than 35 kg/m2
* Significant acute, new onset illness (e.g., flu, gastroenteritis) within two weeks prior to study treatment administration.
* Clinically significant haematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, neurological, or psychiatric disease that may pose a significant safety risk or diminish subject's ability to undergo all study procedures and assessments
* History of immunocompromised status, including a positive HIV (ELISA and Western blot) test result.
* Evidence of active alcohol or drug abuse as indicated by the tests conducted during the screening or baseline evaluations; subject must state they are willing to remain alcohol and drug free for three weeks after study drug administration.
* Use of ASA within 10 days prior to study drug administration.
* Use of Lidocaine, mepivacaine, etidocaine, ropivacaine, and any amide-type anesthetics in any form within 5 elimination half-lives.
* Use of any local anesthetic within 3 days prior to study drug administration.
* Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.
* Any condition that, in the opinion of the Investigator, renders a subject unsuitable for participation in the study. NOTE: A specific rationale must be provided and documented for excluding all prospective subjects deemed unsuitable for the study.

Subjects with Hepatic Impairment:

* Clinically significant abnormal findings other than hepatic impairment.
* Clinical evidence of severe ascites, as judged by the investigator.
* History of surgical portosystemic shunt.
* Fluctuating or rapidly deteriorating hepatic function as indicated by recent history or by widely varying or worsening of clinical and/or laboratory signs of hepatic impairment within the screening period.
* On active Hepatitis treatment with Interferon or other excluded medications (see Appendix 4)

Control Subjects with Normal Hepatic Function:

* Prohibited prescription medications within 14 days prior to dosing; see Appendix 4 for specific medications.
* History or presence of liver disease or liver injury as indicated by an abnormal liver function profile such as SGOT, SGPT, GGT, alkaline phosphatase, or serum bilirubin.
* Hepatitis B as indicated by positive HBs Ag, or Hepatitis C as indicated by positive anti-HCV result.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Serum plasma concentration of SKY0402 | Multiple through 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Janusz Rupinski, Study Director — Pharm-Olam International Polska
Locations (1):
- MTZ Clinical Research, Warsaw, Poland